CLINICAL TRIAL: NCT07033585
Title: Generic Drugs (Dapagliflozin and Saxagliptin) Treat Type 2 Diabetes Patients With Controlled Cancers
Acronym: GD-T2D
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Han Xu, M.D., Ph.D., FAPCR, Sponsor-Investigator, IRB Chair (Industry)
Collaborators: UnitedHealthcare (Other)
Responsible Party: Sponsor-Investigator, Han Xu, M.D., Ph.D., FAPCR, Sponsor-Investigator, IRB Chair, M.D., Ph.D., FAPCR, Sponsor-Investigator, Medical Director, IORG Director, Medical Monitor, Safety Officer, IRB Chair, Medicine Invention Design, Inc
Organization: Medicine Invention Design, Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: ANDA219975 + ANDA220011; NPI-1831468511 (Registry Identifier: HHS, Health Care Provider Individual); NPI-1023387701 (Registry Identifier: HHS, Health Care Provider Organization); FWA00015357 (Registry Identifier: HHS, Human Protections Administrator); IORG0007849 (Registry Identifier: HHS, IORG); IRB00009424 (Registry Identifier: HHS, IRB); ANDA219975 (Registry Identifier: FDA, ANDA); ANDA220011 (Registry Identifier: FDA, ANDA)
Record Dates: First submitted 2025-06-16; First posted 2025-06-24 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Type 2 Diabetes
Keywords: Diabetes; Dapagliflozin; Saxagliptin; Metformin
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — dapagliflozin; saxagliptin

STUDY DESIGN:
Intervention Model Description: * The usual approach group - 300 double blind random group
  * The study approach group - 300 double blind random group
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: No-placebo and random and double blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Farxiga® (dapagliflozin) 10 mg, Onglyza® (saxagliptin) 5 mg, Metformin 500 mg, Oral Mix (Experimental): Farxiga® (dapagliflozin) 10 mg, Onglyza® (saxagliptin) 5 mg, Metformin 500 mg, Oral Mix Prescription
  Interventions: Drug: Farxiga® (dapagliflozin) + Onglyza® (saxagliptin) + Metformin Oral Mix Treat type 2 diabetes
- China Import (dapagliflozin) 10 mg, China Import (saxagliptin) 5 mg, Metformin 500 mg, Oral Mix (Experimental): China Import (dapagliflozin) 10 mg, China Import (saxagliptin) 5 mg, Metformin 500 mg, Oral Mix Prescription
  Interventions: Drug: China Import (dapagliflozin) + China Import (saxagliptin) + Metformin Oral Mix Treat type 2 diabetes

INTERVENTIONS:
Drug: Farxiga® (dapagliflozin) + Onglyza® (saxagliptin) + Metformin Oral Mix Treat type 2 diabetes — Farxiga® (dapagliflozin) 10 mg, Onglyza® (saxagliptin) 5 mg, Metformin 500 mg, Oral Mix Prescription Treat type 2 diabetes patients with controlled cancers
  Other Names: The usual approach group Oral Mix Treat type 2 diabetes
  Arms: Farxiga® (dapagliflozin) 10 mg, Onglyza® (saxagliptin) 5 mg, Metformin 500 mg, Oral Mix
Drug: China Import (dapagliflozin) + China Import (saxagliptin) + Metformin Oral Mix Treat type 2 diabetes — China Import (dapagliflozin) 10 mg, China Import (saxagliptin) 5 mg, Metformin 500 mg, Oral Mix Prescription Treat type 2 diabetes patients with controlled cancers
  Other Names: The study approach group Oral Mix Treat type 2 diabetes
  Arms: China Import (dapagliflozin) 10 mg, China Import (saxagliptin) 5 mg, Metformin 500 mg, Oral Mix

SUMMARY:
Use Dapagliflozin 10 mg, Saxagliptin 5 mg, Metformin 500 mg treat type 2 diabetes patients with controlled cancers

DETAILED DESCRIPTION:
The usual approach group, Farxiga® (dapagliflozin) 10 mg, Onglyza® (saxagliptin) 5 mg, Metformin 500 mg, Oral, 300 double blind random group type 2 diabetes patients with controlled cancers

The study approach group, China Import (dapagliflozin) 10 mg, China Import (saxagliptin) 5 mg, Metformin 500 mg, Oral, 300 double blind random group type 2 diabetes patients with controlled cancers

* Detect Hemoglobin A1c (HbA1c)
* Detect fasting blood glucose (FBG)
* Detect 2-hour postprandial blood glucose (2 hPBG)
* Detect fasting insulin (FINS)
* Detect 2-hour postprandial insulin (2 hPINS)

ELIGIBILITY:
* Select 600 type 2 diabetes patients with controlled cancers.
* Dosage Duration at least 90 days

Inclusion Criteria:

* 1. Clinical diagnosis of type 2 diabetes
* 2. Controlled cancers
* 3. Suitable for enough blood-drawing
* 4. Random and double blind
* 5. Measurable disease
* 6. Adequate organ functions
* 7. Adequate performance status
* 8. Age 24 years old and over
* 9. Sign an informed consent form
* 10. Receive blood-drawing

Exclusion Criteria:

* 1. Uncontrolled cancers
* 2. Pregnancy
* 3. Breast-feeding
* 4. The patients with other serious intercurrent illness or infectious diseases
* 5. The participating patients have serious side effects.
* 6. Serious Allergy to Drugs
* 7. Thrombus or Bleed Tendency
* 8. Serious Risks or Serious Adverse Events of the drug product
* 9. The prohibition of drug products
* 10. Have no therapeutic effects

Ages: 24 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 600 (Estimated)
Dates: Start 2025-06-15 (Actual); Primary Completion 2026-10-18 (Estimated); Study Completion 2026-11-28 (Estimated)

PRIMARY OUTCOMES:
Detect Hemoglobin A1c (HbA1c) | Duration up to 90 days
  Draw blood Detect Hemoglobin A1c (HbA1c)
Detect fasting blood glucose (FBG) | Duration up to 90 days
  Draw blood Detect fasting blood glucose (FBG)
Detect 2-hour postprandial blood glucose (2 hPBG) | Duration up to 90 days
  Draw blood Detect 2-hour postprandial blood glucose (2 hPBG)
Detect fasting insulin (FINS) | Duration up to 90 days
  Draw blood Detect fasting insulin (FINS)
Detect 2-hour postprandial insulin (2 hPINS) | Duration up to 90 days
  Draw blood Detect 2-hour postprandial insulin (2 hPINS)

CONTACTS AND LOCATIONS:
Overall Officials: HAN ID XU, MD/PhD/FAPCR, Study Chair — Medicine Invention Design, Inc. - IORG0007849 - NPI-1023387701; HAN ID XU, MD/PhD/FAPCR, Study Director — Medicine Invention Design, Inc. - IORG0007849 - NPI-1023387701; HAN ID XU, MD/PhD/FAPCR, Principal Investigator — Medicine Invention Design, Inc. - IORG0007849 - NPI-1023387701
Locations (1):
- Medicine Invention Design, Inc. - IORG0007849 - NPI-1023387701, Rockville, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Xu Y, Wu P, Wen W, Chen H. [Short-term intensive combined therapy with metformin, sagliptin and dapagliflozin for newly diagnosed type 2 diabetes: efficacy, weight control and safety]. Nan Fang Yi Ke Da Xue Xue Bao. 2019 Nov 30;39(11):1305-1311. doi: 10.12122/j.issn.1673-4254.2019.11.07. Chinese. PMID 31852646
- See also: FWA < 00015357 > < Medicine Invention Design Incorporation > — http://ohrp.cit.nih.gov/search
- See also: IRB < 00009424 > < Medicine Invention Design Incorporation > — http://ohrp.cit.nih.gov/search
- See also: IORG < 0007849 > < Medicine Invention Design Incorporation > — http://ohrp.cit.nih.gov/search

DOCUMENTS (3):
  • Study Protocol (2025-06-16): https://cdn.clinicaltrials.gov/large-docs/85/NCT07033585/Prot_000.pdf
  • Statistical Analysis Plan (2025-06-16): https://cdn.clinicaltrials.gov/large-docs/85/NCT07033585/SAP_001.pdf
  • Informed Consent Form (2025-06-16): https://cdn.clinicaltrials.gov/large-docs/85/NCT07033585/ICF_002.pdf